CLINICAL TRIAL: NCT02650739
Title: Duration of Prone Positioning After Macular Hole Surgery Determined by Swept Source Optical Coherence Tomography
Brief Title: Optical Coherence Tomography-based Positioning for Macular Hole Surgery
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Professor of Ophthalmology, Kyorin University
Other Study IDs: Kyorineye0021
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Macular Hole Surgery
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SS-OCTdetermined group: Eyes with macular hole surgery that the postoperative prone positioning was discontinued after detecting a closure by SS-OCT
  Interventions: Procedure: Macular hole surgery
- Control group: Eyes with macular hole surgery that the halting of the prone position was determined by the surgeon
  Interventions: Procedure: Macular hole surgery

INTERVENTIONS:
Procedure: Macular hole surgery — Vitrectomy with internal limiting membrane removal and gas tamponade
  Other Names: Vitrectomy

SUMMARY:
The efficacy of macular hole (MH) surgery with the halting of prone positioning by monitoring the MH closure in the swept source optical coherence tomographic (SS-OCT) images was compared with the surgery by the surgeon's decision. The macular hole closure and visual outcome were compared.

DETAILED DESCRIPTION:
The efficacy of macular hole (MH) surgery with the halting of prone positioning by monitoring the MH closure in the swept source optical coherence tomographic (SS-OCT) images was compared with the surgery by the surgeon's decision. All eyes were treated by pars plana vitrectomy, internal limiting membrane peeling, and gas tamponade. MH closure was defined as a connection of the edges of the sensory retina in the SS-OCT images.The macular hole closure and visual outcome were compared.

ELIGIBILITY:
Inclusion Criteria:

* The patients were followed more than 2 months.

Exclusion Criteria:

* Eye with axial length more than 26.0 mm

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The efficacy of macular hole (MH) surgery with the halting of prone positioning by monitoring the MH closure in the swept source optical coherence tomographic (SS-OCT) images in 60 eyes was compared with the 69 eyes with same surgical procedure but the prone position determined by the surgeon's decision.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Macular hole closure | Changes from baseline to 1, 2 months
  Closure of macular hole

SECONDARY OUTCOMES:
Visual acuity before and after surgery | Changes from baseline to 1, 2 months
  Vision

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center

IPD SHARING:
Plan to Share IPD: No